CLINICAL TRIAL: NCT06849141
Title: The Effect of the Role Performance Strengthening Program Based on the Roy Adaptation Model on the Adaptive Performance and Competence of Nurses Working in Pandemic Units
Brief Title: The Effect of the Role Performance Strengthening Program on the Adaptive Performance and Competence of Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: Akdeniz University Hospital (Other)
Responsible Party: Principal Investigator, Belkıs Simsek, PhD, Akdeniz University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KAEK-751
Record Dates: First submitted 2025-02-11; First posted 2025-02-27 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Adaptation; Competence; Psychiatric Nursing; Psychoeducation; Mixed Method Implementation Study
Keywords: psychiatric nursing; psychoeducation; role performance; Roy Adaptation Model; coronavirus pandemic

STUDY DESIGN:
Intervention Model Description: The research process has four stages: Pre-action, action, post-action and follow-up. In the Pre-Action Stage, quantitative data were collected from 54 nurses volunteered to participate in the research. According to the obtained score averages determined a risk group. This risk group consisted of 42 nurse. 35 of these nurses accepted to have a semi-structured interview before the action. With the information obtained from the analysis of the collected quantitative and qualitative data, the "Role Performance Strengthening Program" was structured based on the Roy Adaptation Model. In the Action Stage, 35 nurses were invited to participate in the RPSP, and 10 nurses accepted to participate. A psychoeducation program was implemented to 10 nurses. In the Post-Action Stage, quantitative and qualitative measurements were repeated one week after the last session with each nurse. In the Follow-up Stage, quantitative and qualitative measurements were repeated four weeks after the last sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nurses who were implemented the "Role Performance Strenghthening Program (RPSP)" (Experimental): Within the scope of the doctoral thesis study, the "Role Performance Enhancement Program (RPGP), an individual psychoeducation program produced within the framework of cognitive behavioral approach elements and based on the Roy Adaptation Model, was applied to 10 nurses. Each nurse was worked with individually. Sessions were conducted online or face-to-face, at the time and place preferred by the nurses, once a week. The program consisted of 6 sessions. Each session lasted 45-90 minutes on average. However, the duration of each session could be extended according to the needs of the nurses. After the application, post-action measurements were made one week later and follow-up measurements were made four weeks later.
  Interventions: Other: Role Performance Strenghthening Program

INTERVENTIONS:
Other: Role Performance Strenghthening Program — This intervention was developed by the researcher within the scope of her doctoral dissertation. The intervention is an individual psychoeducation program; it was written and structured within the framework of cognitive behavioral therapy, based on the Roy Adaptation Model. The intervention was structured on the idea of empowering nurses working in pandemic units.

SUMMARY:
The "Role Performance Strenghthening Program (RPSP)" based on the Roy Adaptation Model was structured to increase the competence and adaptive performance levels of nurses working in pandemic units and to strenghthen role performance of nurses. In the measurements made after the completion of the program, it was determined that the competence and adaptive performance level of the nurses increased. It was found that the Roy Adaptation Model was suitable for use in research to be conducted on a nurse sample regarding coping with the challenges caused by coronavirus pandemic. It is recommended that the RPSP be included in institutional training programs.

DETAILED DESCRIPTION:
It has been understood that supporting the mental health and resilience of nurses who are vulnerable to the difficulties experienced during the pandemic process is of great importance. In this context, it has been revealed that there is a need for supportive psychiatric nursing practices; that psychiatric nurses need to help their colleagues cope with difficulties during difficult processes such as the pandemic. Based on this need, a psychoeducation program was written in this doctoral thesis to support and strengthen nurses during the pandemic process. This program, called "Role Performance Strengthening Program", is shaped within the framework of cognitive behavioral approach elements and is based on the Roy Adaptation Model. It is thought that the competence and adaptive performance level of nurses will increase through this structured psychoeducation program; therefore, the competence and adaptive performance level of nurses will be maintained and even increased during difficult processes such as the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Working as a nurse in pandemic clinics, pandemic intensive care units or the orange area of the emergency room,
* Having a competency score average below 26 as a result of measurements made with the Nursing Competency Scale,
* Accepting to participate in the research in writing and verbally,
* Accepting to participate in all sessions of the Role Performance Strenghthening Program. -

Exclusion Criteria:

• It has been determined that the person is continuing a therapy program to cope with the problems he/she experiences due to working during the pandemic. -

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-04-17 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Scoring below 26 on the "Nurse Competence Scale" | All quantitative and qualitative data of the first phase of the research were collected in approximately 8 weeks.
  Quantitative data collection forms were first given to 54 nurses by the researcher and collected. After the scores obtained from these forms were collected and averaged, 42 nurses who received less than 26 points from the Nurse Competence Scale were selected. Getting less than 25 points from the Nurse Competence Scale is an indicator of low level of competence.
  Nurses' competence levels were measured with a visual analog scale (VAS) ranging from 0 to 100 points. Scores below 25 indicate "low competence"; scores between 25 and 49 indicate "slightly good competence"; scores between 50 and 75 indicate "good competence"; and scores above 75 indicate "very good competence".

CONTACTS AND LOCATIONS:
Overall Officials: İlhan Günbayı, Prof. Dr., Study Director — Akdeniz University Faculty of Education, Department of Educational Sciences
Locations (1):
- Akdeniz University Hospital, Antalya, Konyaalti, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yilmaz A, Seren Intepeler S. Opinions of emergency nurses in Turkey on their work environment during the COVID-19 pandemic and its relationship with their health: A qualitative study. Heliyon. 2023 Nov 25;9(12):e22716. doi: 10.1016/j.heliyon.2023.e22716. eCollection 2023 Dec. PMID 38144309
- [Background] Yiğitol B, Büyükmumcu S. Covid-19 Korkusu, Kişilik Özellikleri, İş Performansı ve İşten Ayrılma Niyeti Arasındaki Yordayıcı İlişkilerin İncelenmesi. OPUS International Journal of Society Researches, 2021; 17(Pandemi Özel Sayısı): 3414-3447.
- [Background] Senesac P, Roy C. Callista Roy's Adaptation Model. In: Smith, MC, Gullett, DL. eds. Nursing Theories & Nursing Practice. 5thed. Philadelphia: FA Davis Company; 2019, Chapter 10, p: 149-164.
- [Background] Savsar A, Damar HT, Aktaş FÖ. Operating Room Nurses' Metaphorical Perceptions of Coronavirus Disease 2019, Quarantine, and Mask Concepts: A Qualitative Study. J Nursology, 2023; 26(3), 167-174.
- [Background] Roy SC. The Roy Adaptation Model (3rd Ed.) New Jersey: Pearson Education & Upper Saddle River; 2009(b).
- [Background] Roy SC. Elements of the Roy Adaptation Model. In: Roy SC, ed. The Roy Adaptation Model. 3rd ed. New Jersey: Pearson Education; 2009(a).
- [Background] Roy C. Spiritualty based on the Roy adaptation model for use in practice, teaching and research. Aquichan, 2018; 18(4): 393-394.
- [Background] Roy C. Research based on the Roy adaptation model: last 25 years. Nurs Sci Q. 2011 Oct;24(4):312-20. doi: 10.1177/0894318411419218. PMID 21975478
- [Background] Roy C. Extending the Roy adaptation model to meet changing global needs. Nurs Sci Q. 2011 Oct;24(4):345-51. doi: 10.1177/0894318411419210. PMID 21975483
- [Background] Roy C. A theorist envisions the future and speaks to nursing administrators. Nurs Adm Q. 2000 Winter;24(2):1-12. doi: 10.1097/00006216-200001000-00004. PMID 10765251
- [Background] Roy C, Zhan L. Sister Callista Roy's Adaptation Model and Its Applications. (Chapter 17). Nursing Theories and Nursing Practice. 2. Edition. F.A. Davis Company; 2006.
- [Background] Pulakos ED, Schmitt N, Dorsey DW, Arad S, Borman WC, Hedge JW. Predicting adaptive performance: Further tests of a model of adaptability. Hum perform, 2002; 15(4): 299-323.
- [Background] Pulakos ED, Dorsey DW, White SS. Adaptability in the workplace: Selecting an adaptive workforce. In Understanding adaptability: A prerequisite for effective performance within complex environments. Emerald Group Publishing Limited; 2006.
- [Background] Mensinger JL, Brom H, Havens DS, Costello A, D'Annunzio C, Durning JD, Bradley PK, Copel L, Maldonado L, Smeltzer S, Yost J, Kaufmann P. Psychological responses of hospital-based nurses working during the COVID-19 pandemic in the United States: A cross-sectional study. Appl Nurs Res. 2022 Feb;63:151517. doi: 10.1016/j.apnr.2021.151517. Epub 2021 Oct 27. PMID 35034708
- [Background] Menard AD, Soucie K, Ralph J, Chang YY, Morassutti O, Foulon A, Jones M, Desjardins L, Freeman L. One-year follow-up of hospital nurses' work experiences during the COVID-19 pandemic: A qualitative study. J Adv Nurs. 2023 Jul;79(7):2502-2513. doi: 10.1111/jan.15599. Epub 2023 Feb 24. PMID 36825468
- [Background] Masters K. Roy Adaptation Model: Sister Callista Roy. In: Nursing Theories: A Framework for Professional Practice. 2nd ed. Burlington: Jones & Barlett Learning; 2015.
- [Background] Hannon-Engel SL. Knowledge development: the roy adaptation model and bulimia nervosa. Nurs Sci Q. 2008 Apr;21(2):126-32. doi: 10.1177/0894318408315015. PMID 18378822
- [Background] Gunbayi I. Rigor in qualitative research. JAQMER, 2024; 3(2), 1-7.
- [Background] Gunbayi I. Knowledge-constitutive interests and social paradigms in guiding mixed methods research (MMR). JOMES, 2020(b); (1), 44-56.
- [Background] Gunbayi I. Action Research as a Mixed Methods Research: Definition, Philosophy, Types, Process, Political and Ethical Issues and Pros and Cons. JOMES, 2020(a); 2: 16-25.
- [Background] Guba EG. Criteria for assessing the trustworthiness of naturalistic inquiries. Educational Communication and Technology Journal 1981; 29(2), 75-91.
- [Background] Fawcett J. Using the Roy adaptation model to guide research and/or practice: construction of Conceptual-Theoretical-Empirical systems of knowledge. Aquichan, 2009; 9(3), 297-306.
- [Background] Tsukuda M, Kayano T, Ito Y. Experiences of COVID-19-Related Stigma: A Qualitative Study on Nurses Caring for Patients With COVID-19. J Nurs Res. 2022 Dec 1;30(6):e241. doi: 10.1097/jnr.0000000000000528. PMID 36302148
- [Background] Takase M, Yamamoto M, Sato Y. The factors related to self-other agreement/disagreement in nursing competence assessment: Comparative and correlational study. Int J Nurs Stud. 2018 Apr;80:147-154. doi: 10.1016/j.ijnurstu.2018.01.011. Epub 2018 Feb 2. PMID 29426015
- [Background] Takase M, Teraoka S. Development of the Holistic Nursing Competence Scale. Nurs Health Sci. 2011 Dec;13(4):396-403. doi: 10.1111/j.1442-2018.2011.00631.x. Epub 2011 Aug 31. PMID 21883769
- [Background] Roy C. Adversity and theory: the broad picture. Nurs Sci Q. 2008 Apr;21(2):138-9. doi: 10.1177/0894318408316407. No abstract available. PMID 19023928
- [Background] Pulakos ED, Arad S, Donovan MA, Plamondon KE. Adaptability in the workplace: development of a taxonomy of adaptive performance. J Appl Psychol. 2000 Aug;85(4):612-24. doi: 10.1037/0021-9010.85.4.612. PMID 10948805
- [Background] MacKay MM, Powers K, Jordan K. The COVid-19 pandemic through the eyes of pediatric nurses: A qualitative study. J Pediatr Nurs. 2023 Jan-Feb;68:52-59. doi: 10.1016/j.pedn.2022.09.015. Epub 2022 Nov 7. PMID 36357232
- [Background] Littzen-Brown C, Dolan H, Norton A, Bethel C, May J, Rainbow J. Unbearable suffering while working as a nurse during the COVID-19 pandemic: A qualitative descriptive study. Int J Nurs Stud Adv. 2023 Dec;5:100127. doi: 10.1016/j.ijnsa.2023.100127. Epub 2023 Apr 12. PMID 37082653
- [Background] Fukada M. Nursing Competency: Definition, Structure and Development. Yonago Acta Med. 2018 Mar 28;61(1):1-7. doi: 10.33160/yam.2018.03.001. eCollection 2018 Mar. PMID 29599616
- [Background] Fawcett J. Thoughts About the Metaparadigm of Nursing: Contemporary Status and Recommendations for Evolution. Nurs Sci Q. 2023 Jul;36(3):303-305. doi: 10.1177/08943184231169770. PMID 37309143
- [Background] Fawcett J. The metaparadigm of nursing: present status and future refinements. Image J Nurs Sch. 1984 Summer;16(3):84-9. doi: 10.1111/j.1547-5069.1984.tb01393.x. No abstract available. PMID 6565629
- [Background] Fawcett J. More Thoughts About the Evolution of the Metaparadigm of Nursing: Addition of Culture as Another Metaparadigm Concept and Definitions of All the Concepts. Nurs Sci Q. 2024 Apr;37(2):183-184. doi: 10.1177/08943184231224409. PMID 38491881
- [Background] Fawcett J. Contemporary nursing knowledge analysis and evaluation of nursing models and theories. Fa Davis comp. USA; 2006.
- [Background] Fawcett J, Desanto-Madeya S. Contemporary nursing knowledge: Analysis and evaluation of nursing models and theories. FA Davis; 2012.
- See also: ICN COVID-19 Update: Occupational risks to nurses must be minimised to enable them to continue their vital work — https://www.icn.ch/sites/default/files/inline-files/PR_10_COVID-19%20update%20-%2020%20March%202020.pdf
- See also: Guidelines on mental health nursing. — https://www.icn.ch/sites/default/files/2024-07/ICN_MentalHealthNursingGuidelines-2024_EN_web.pdf